CLINICAL TRIAL: NCT02134275
Title: Whole Body Vibration Training for Healthy Body Composition in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kerri Winters, Research Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10504
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Obesity; Weight Gain
Keywords: whole body vibration training; young adult; weight gain; obesity; randomized clinical trial
MeSH Terms: conditions — Obesity; Weight Gain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole body vibration training (Experimental): Whole body vibration training (timed stand on vibration platform) 3 20-minute sessions per week for 6 months
  Interventions: Behavioral: Whole body vibration training
- Control group (Placebo Comparator): No significant changes to diet, exercise and lifestyle.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Whole body vibration training — Each whole body vibration session will consist of a 20 min timed stand on the vibration platform where participants will stand with their knees in a slightly flexed position (120°) while the plate oscillates. The vibration frequency will be set at ranges between 20-40Hz and the amplitude set at 2mm displacement.
  Arms: Whole body vibration training
Behavioral: Control group — Participants in this group will be asked to not make any significant changes to their lifestyle behaviors, such as diet and exercise, for the duration of the study.
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the benefits and feasibility of a whole body vibration (WBV) exercise program as a method of preventing weight gain in young adults.

ELIGIBILITY:
Inclusion Criteria:

1. BMI that is between 22-29.9 kg/m2
2. History of being weight stable (± 2 kg) for three months prior to beginning the intervention
3. Not currently on a prescribed diet plan to lose weight and no plan to begin one
4. Not consistently engaged in physical activity that meets current public health recommendations of 150 minutes of moderate to vigorous physical activity in the previous 6 months
5. Currently enrolled as an undergraduate student in a degree-granting college or university
6. Planning to reside in the Portland Metro area for the duration of the study

Exclusion Criteria:

1. Health condition that would prevent participation in moderate intensity physical activity program.
2. For female participants, pregnancy or plans to become pregnant during the study period (source documentation: self-report on HHQ)
3. Currently smoking/tobacco products or initiation of smoking/tobacco during the study
4. Alcohol consumption exceeding 3 drinks per day or a total of 18 drinks per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in body composition (total body mass, fat-free mass, fat mass, regional fat mass, android/gynoid ratio and % body fat) across baseline, 3 and 6 months | baseline, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU School of Nursing, Portland, Oregon, United States